CLINICAL TRIAL: NCT04444427
Title: An Open-Label, Multicenter, Phase 1b/2 Study to Establish Safety, Tolerability, and Optimal Dosing Strategy of GLR2007 in Subjects With Advanced Solid Tumors
Brief Title: Evaluation of GLR2007 for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GLP-CDK-1009
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-07

CONDITIONS: Non-small Cell Lung Cancer; Glioblastoma Multiforme
Keywords: Non-small Cell Lung Cancer; Glioblastoma Multiforme; Breast Cancer; Advanced Solid Tumors; GLR2007
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Glioblastoma; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Part 1 employs a dose-escalation design to determine the recommended phase 2 dose. This is followed by Part 2, which involves parallel dosing of 3 different cohorts at the dose determined in Part 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation (Experimental): Dose escalation cohorts are planned to determine the maximum tolerated dose or recommended phase 2 dose of GLR-2007, as well as expansion cohorts and a Phase 2 cohort.
  Interventions: Drug: GLR2007
- Part 2: Dose Expansion - Cohort A (Experimental): Participants who have received 2 or more second-line therapies, with at least 1 line of standard therapy, for their non-small cell lung cancer (NSCLC) will be dosed the maximal tolerated dose of GLR2007 as determined in Part 1 until lack of tolerance or disease progression.
  Interventions: Drug: GLR2007
- Part 2: Dose Expansion - Cohort B (Experimental): Participants who have received 2 or more second-line therapies, with at least 1 line of standard therapy, for their brain metastases of breast or NSCLC origin will be dosed the maximal tolerated dose of GLR2007 as determined in Part 1 until lack of tolerance or disease progression.
  Interventions: Drug: GLR2007
- Part 2: Dose Expansion - Cohort C (Experimental): Participants experiencing their first recurrence glioblastoma multiforme (GBM) will be dosed the maximal tolerated dose of GLR2007 as determined in Part 1 until lack of tolerance or disease progression.
  Interventions: Drug: GLR2007

INTERVENTIONS:
Drug: GLR2007 — Administered orally, once daily for 21 days followed by a 7-day treatment holiday.
  Other Names: GLR2007-237FA

SUMMARY:
Evaluation of GLR2007 for Advanced Solid Tumors

DETAILED DESCRIPTION:
An Open-Label, Multicenter, Phase 1b/2 Study to Establish Safety, Tolerability, and Optimal Dosing Strategy of GLR2007 in Subjects with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. For Part 1 (Dose Escalation): Participants with advanced solid tumors who are refractory or intolerant to therapies known to provide clinical benefit.

   1. For Part 1 (Dose Escalation): The participant must have histological or cytological evidence of cancer (a solid tumor) that is advanced and/or metastatic. Biopsy is allowed by protocol if no histology or cytology records are available.
   2. For Part 2 (Dose Expansion): The participant must have histological or cytological evidence of cancer that is advanced and/or metastatic.
2. For Part 1 (Dose Escalation): The participant has measurable or non-measurable disease.
3. For Part 2 (Dose Expansion): The participant has measurable disease.
4. The participant has given written informed consent prior to all study-specific procedures.
5. The participant has adequate hematologic, hepatic, and renal function.
6. The participant has discontinued all prior cancer therapies (including chemotherapy, immunotherapy, and investigational therapy) for at least 21 days for myelosuppressive agents or 14 days for radiotherapy and non-myelosuppressive agents, prior to receiving GLR2007, and has recovered from the acute effects of therapy (treatment related toxicity resolved to ≤Grade 1) except for residual alopecia.
7. The participant is willing and able to make themselves available for the duration of the study and is willing and able to follow study procedures.
8. The participant meets contraceptive requirements.
9. The participant has an estimated life expectancy of ≥3 months.
10. The participant agrees to minimize ultraviolet exposure and sunlight for the duration of their study participation.
11. A diagnostic contrast-enhanced magnetic resonance imaging (MRI) of the brain must be performed within 28 days prior to registration. Contrast-enhanced computed tomography (CT) is acceptable if MRI is not possible.

Cohort-specific inclusion criteria Part 2 (Cohort A, NSCLC)

1. Histologically or cytologically confirmed NSCLC.
2. Participants must have received at least 1 line of standard therapy for metastatic disease, including platinum-based chemotherapy and an immune checkpoint inhibitor given together or as separate lines of therapy, unless participants are ineligible for or cannot tolerate such therapy.
3. Participants with anaplastic lymphoma kinase (ALK), epidermal growth factor receptor (EGFR), proto-oncogene tyrosine-protein kinase ROS (ROS1), v-Raf murine sarcoma viral oncogene homolog B (BRAF), and neurotrophic receptor tyrosine kinase 1 (NTRK) aberrations must have received therapy directed at their molecular aberration in order to enroll on this study.

Part 2 (Cohort B, Brain metastases of breast or NSCLC origin)

1. Histologically or cytologically confirmed NSCLC or breast cancer at primary site.
2. Participants with inoperable brain metastases (prior radiation therapy and/or stereotactic radiosurgery is allowed). A neurosurgical consult is at the discretion of the investigator.
3. Participants with brain metastases of NSCLC origin must have received at least 1 line of standard therapy for metastatic disease, including platinum-based chemotherapy and an immune checkpoint inhibitor given together or as separate lines of therapy, unless participants are ineligible for or cannot tolerate such therapy.
4. Participants with ALK, EGFR, ROS1, BRAF, and NTRK aberrations must have received therapy directed at their molecular aberration in order to enroll on this study.
5. Participants with brain metastases from breast cancer who have previously received CDK4/6 inhibitors.

Part 2 (Cohort C, GBM)

1. Histologically confirmed diagnosis of a recurrent primary World Health Organization Grade IV malignant glioblastoma. Participants with recurrent disease whose diagnostic pathology confirmed glioblastoma will not need re-biopsy. Participants with prior low-grade glioma or anaplastic glioma are eligible if histologic assessment demonstrates transformation to GBM.
2. First recurrence of GBM.
3. Candidate for surgical partial or gross-total resection.
4. Radiographic demonstration of disease progression by contrast-enhanced CT or MRI following prior therapy.
5. At least 2 weeks between prior surgical resection and adequate wound healing.
6. At least 12 weeks from prior radiotherapy unless there is either histopathologic confirmation of recurrent tumor or new enhancement on MRI outside of the treatment field.

Exclusion Criteria:

1. The participant has a personal history of any of the following conditions: major surgical resection involving the stomach or small bowel recurrent, unexplained or cardiac-related syncopal episodes within the last 6 months or ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation).
2. Any concurrent malignancies currently requiring treatment or for which treatment would be deemed necessary within 3 months of enrollment; prostate cancer with androgen deprivation therapy, basal cell cancer, and squamous cell cancers are allowed.
3. The participant is pregnant or lactating.
4. The participant is immunocompromised and known to be human immunodeficiency virus positive. The participant has an active bacterial, fungal, and/or known viral infection (for example, hepatitis B surface antigen or hepatitis C antibodies).

Cohort-specific exclusion criteria:

Part 2 (Cohort A, NSCLC): The participant has NSCLC with worsening symptoms within 14 days prior to receiving GLR2007.

Part 2 (Cohort B, Brain metastases of breast or NSCLC origin): The participant has CNS metastasis with worsening symptoms within 14 days prior to receiving GLR2007.

Part 2 (Cohort C, GBM): The participant has GBM with worsening symptoms within 14 days prior to receiving GLR2007.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Dose-limiting Toxicities | Up to 12 Months
Dose Escalation: Incidence And Severity Of Adverse Events, Including The Incidence Of Dose-limiting Toxicities Within The First Cycle | Up to 12 Months
Dose Expansion: Incidence And Severity Of Adverse Events | Up to 96 Weeks

SECONDARY OUTCOMES:
Dose Escalation: Objective Response Rate | 8 Weeks
  Defined by response evaluation criteria in solid tumors (RECIST) Version 1.1 (solid tumors) or by response assessment in neuro-oncology (RANO) (brain metastases and GBM).
Dose Expansion: Objective Response Rate | 12, 24, 36, 48, 60, 72, 84, and 96 Weeks
  Defined by RECIST Version 1.1 or by RANO as appropriate.
Dose Escalation And Expansion: Maximum Observed Plasma Concentration After Single And Multiple Oral Dose Administrations | 0, 0.25, 0.5, 1, 2, 4, 6, 8, and 24 hours postdose
Dose Escalation And Expansion: Time At Which Maximum Plasma Concentration Is Observed And Apparent Half-life After Single And Multiple Oral Dose Administrations | 0, 0.25, 0.5, 1, 2, 4, 6, 8, and 24 hours postdose
Dose Escalation And Expansion: Area Under The Plasma Concentration-time Curve From 0 To Last Measurable Concentration And From 0 To Infinity After Single And Multiple Oral Dose Administrations | 0, 0.25, 0.5, 1, 2, 4, 6, 8, and 24 hours postdose
Dose Escalation And Expansion: Accumulation Ratio After Single And Multiple Oral Dose Administrations | 0, 0.25, 0.5, 1, 2, 4, 6, 8, and 24 hours postdose
Dose Escalation And Expansion: Steady-state Volume Of Distribution After Single And Multiple Oral Dose Administrations | 0, 0.25, 0.5, 1, 2, 4, 6, 8, and 24 hours postdose
Dose Escalation And Expansion: Clearance After Single And Multiple Oral Dose Administrations | 0, 0.25, 0.5, 1, 2, 4, 6, 8, and 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Lazaroff, MSN, Study Director — Gan and Lee Pharmaceuticals, USA Corp
Locations (4):
- United States (4):
  - USA002, Lafayette, Indiana
  - USA005, Omaha, Nebraska
  - USA001, Philadelphia, Pennsylvania
  - USA004, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No